CLINICAL TRIAL: NCT00662207
Title: Two Devices for Reflex Voiding Following SCI: Urodynamic Evaluation
Brief Title: Two Devices for Reflex Voiding Following Spinal Cord Injury
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: B6176-R
Record Dates: First submitted 2008-04-01; First posted 2008-04-21 (Estimated); Results first posted 2014-11-05 (Estimated); Last update posted 2014-11-05 (Estimated); Status verified 2014-11

CONDITIONS: Spinal Cord Injury; Urinary Incontinence
Keywords: electric stimulation; urethral obstruction; urodynamics; urology
MeSH Terms: conditions — Spinal Cord Injuries; Urinary Incontinence; Urethral Obstruction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental): Use a vibrator on the patient's bottom to determine if it will induce a bladder contraction; Use an anal dilator to determine if urethral relaxation will occur
  Interventions: Device: Vibrator; Procedure: Anal dilator

INTERVENTIONS:
Device: Vibrator — A vibrator will be applied to the patient's bottom to determine if it will induce a bladder contraction
  Other Names: perinuem vibrator
Procedure: Anal dilator — A balloon will be used for anal dilation to determine if it will result in relaxation of the pelvic floor and urethral sphincter. An anal dilator is being conduced with the balloon
  Other Names: Modified rectal balloon for anal dilation

SUMMARY:
The purpose of this investigation is to evaluate methods in spinal cord injured individuals to improve reflex urination. Anal dilation will be investigated to reduce high urethral resistance and a vibrator on the patient's bottom will be tested to induce more sustained bladder contractions for better bladder emptying.

DETAILED DESCRIPTION:
Catheters are often used by individuals emptying their bladder following spinal cord injury. Reflex voiding is one of the bladder emptying methods, and it relies on spontaneous bladder contractions for voiding. These contractions occur with normal bladder filling or can be induced with suprapubic tapping and hair pulling. Poor voiding responses with reflex voiding can occur because of unwanted contractions of the urethra during bladder contractions and/or unsustained bladder contractions that result in high residual urine. The focus of this investigation is methods to reduce the high urethral resistance and to induce more sustained bladder contractions.

Obj.1. Measure pelvic floor contractile activity including the pelvic floor relaxation response (urethral and anal pressures, and EMG and the bulbocavernosus reflex) during dilation of the anus with digits or a balloon for 60 sec at diameters of 2, 3.5 and 5 cm.

Obj. 2. Measure urodynamic parameters (urethral and anal pressures, EMG, urine flow rates and bladder pressure) and compare three somatic methods of inducing bladder contractions, which are vibration (3 mm conducted at 100 strokes per second) at suprapubic and perineum (between the scrotum and anus) locations and tapping/suprapubic hair pulling. Conduct procedures using 80% of cystometric capacity and define a responder to any of the three interventions as an increase of 10 cm H20 pressure or greater. For nonresponders go to objective 4.

Obj. 3. For responders to Ob. 2, further evaluate effects of perineum vibration by conducting comparisons with (1) anal dilation to no dilation; (2) A vibration stroke length of 1.5 mm to 3 mm; (3) A bladder volume of 50% cystometric capacity to 80%.

Obj. 4. Compare the urodynamic responses to spontaneous bladder contractions induced by bladder filling (cystometry) with and without anal dilation.

Obj. 5. Conduct a human factors assessment. Determine problems with use of the current perineum vibration and anal dilation devices. Evaluate if curving the tip of the insertion device for the anal dilator would facilitate insertion and if the use of a plastic bag would improve hygiene. Discuss features important for a user-friendly home-use device.

Design & Methods: All objectives will be conducted during a single, urodynamic, testing protocol. Fifteen male SCI patients with upper-motor-neuron injuries will be enrolled. Urodynamic responses are our primary measure. These include urethral and anal sphincter pressures and anal surface EMG, bladder contractions including peak pressure and duration of pressure, voiding responses including peak voiding rate and duration of voiding. These measures will be evaluated during anal dilation and perineum vibration methods alone and in combination. Anal dilation protocols will include random and duplicated testing. Vibration methods will only be done once to limit the risk of autonomic dysreflexia. Analysis of variance followed by Student-Neuman-Keuls post hoc test will be conducted to assess significant differences.

Importance of Findings: Results from these studies will provide evidence for anal dilation to reduce DSD and perineum vibration to improve bladder contractions. Thus, these studies could provide important evidence for improved methods of RV for individuals with SCI. During this pilot study, subjects will not be counseled to conduct RV for their daily or regular bladder management program.

ELIGIBILITY:
Inclusion Criteria:

Male Veterans using Hines VA Hospital SCI Service that have upper motor neuron injuries

Exclusion Criteria:

* Can voluntarily control their urination
* Surgically removed external urethral sphincter in men or replaced bladder
* Any implanted devices in the lower urinary tract
* Female
* Urinary tract infection in the prior 3 months or untreated urinary tract infection, or bladder pathology such as a tumor or stones
* History of autonomic dysreflexia
* Anal inflammation or pathology
* Use of Indwelling (Foley) catheter as the primary method of bladder management; note patients will be included if they only occasionally use a Foley catheters; for example, during traveling
* Not under 18 or over 70 years old and in good health
* Less than 3-months after injury and before the return of bladder reflexes
* Lower motor neuron spinal cord injury
* Not competent to understand the study and the consent and willing to participate in study.

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2008-10; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Walter, PhD, Principal Investigator — Edward Hines Jr. VA Hospital
Locations (1):
- Edward Hines, Jr. VA Hospital, Hines, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Only spinal cord injured (SCI) patients using intermittent catheterization or reflex voiding with upper motor neuron injuries participated in this study. Three SCI male patients were enrolled and no adverse events occurred.
Groups:
- Experimental Group: Use a vibrator on the patient's bottom to determine if it will induce a bladder contraction; or use a dilator of the anus to determine if urethral relaxation will occur
  Vibrator: A vibrator will be applied to the patient's bottom to determine if it will induce a bladder contraction
  Anal dilator: A balloon will be used for anal dilation to determine if it will result in relaxation of the pelvic floor and urethral sphincter
  A single urodynamic testing protocol was conducted for each patient. Techniques included urodynamic catheters, perineum vibration, and anal dilation with a balloon dilator.
  Responses of the bladder and the external urethral and anal sphincters were recorded
Period: Overall Study
Arm/Group | Experimental Group
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: baseline anal pressure
Arm/Group | All Participants
Number analyzed (Participants) | 3
Age, Customized [Number; unit: participants]
  Between 50 and 60 years old | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 3
Number of Participants with Upper-Motor-Neuron Injuries for SCI [Number; unit: participants] | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Change in Bladder Pressure
Description: Measured via pressure catheter in bladder with a pressure transducer
Time Frame: 3 hour recording session
Measure: Number; unit: participants
Arm/Group | Experimental Group
Number analyzed (Participants) | 3
participants | 0

2. Primary Outcome: Number of Participants With a Change in External Urethral Pressure
Description: Measured via balloon catheter
Time Frame: 3 hour recording session
Measure: Number; unit: participants
Arm/Group | Experimental Group
Number analyzed (Participants) | 3
participants | 0

3. Primary Outcome: Number of Participants With a Change in Anal Sphincter Pressure
Description: Measured via balloon catheter
Time Frame: 3 hour recording session
Measure: Number; unit: participants
Arm/Group | Experimental Group
Number analyzed (Participants) | 3
participants | 0

4. Primary Outcome: Number of Participants With a Urethral Sphincter Contractions
Time Frame: 3 hour recording session
Measure: Number; unit: participants
Arm/Group | Experimental Group
Number analyzed (Participants) | 3
participants | 0

ADVERSE EVENTS:
Time Frame: 3 hour recording session
Arm/Group | Experimental Group
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes